CLINICAL TRIAL: NCT01568710
Title: Measurement of the Reactive Hyperemia Index in Sickle Cell Patients During Pain Crisis and After Recovery
Brief Title: Blood Flow and Pain Crises in People With Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120101; 12-H-0101
Record Dates: First submitted 2012-03-30; First posted 2012-04-02 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10-05

CONDITIONS: Sickle Cell Disease
Keywords: Blood Flow; Endothelium; Nitric Oxide; Oximetry; Laser Doppler; Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Many people with sickle cell disease have repeated episodes of severe pain that lasts for days, requiring hospital care. These episodes, called pain crises, may be caused by changes in blood flow. Researchers want to study blood flow in people with sickle cell disease who are having a pain crisis and compare it with their blood flow after the pain crisis has resolved. They also want to compare these measurements against blood flow in healthy people who do not have sickle cell disease.

Objectives:

- To study whether changes in blood flow cause pain crises in people with sickle cell disease.

Eligibility:

* Individuals at least 18 years of age who have sickle cell disease and are being treated for a pain crisis.
* Individuals at least 18 years of age who have sickle cell disease and are not experiencing a pain crisis.
* Healthy volunteers matched by age and gender with the participants who have sickle cell disease.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected.
* Participants having a sickle cell pain crisis will have two visits, one during the crisis and one about 4 weeks after the crisis has resolved.
* Participants not having a sickle cell pain crisis will have one or two study visits. Blood samples will be collected during at least one of these visits.
* Healthy volunteers will have one or two study visits. Blood samples will be collected during at least one of these visits.
* During each visit for all participants, cameras and blood flow monitoring equipment will be used to measure blood flow in the forearm.

sickle cell disease.

DETAILED DESCRIPTION:
Severe recurrent pain is the most common cause of acute morbidity in sickle cell disease1. The underlying pathogenesis was initially thought to be ischemia from obstruction of capillary beds by stiffened red blood cells; however, there is evidence that other factors contribute to the pathogenesis of sickle cell pain crisis, such as inflammation and coagulation, ischemia-reperfusion injury, angiogenesis balance, and vasomotor tone processes that are regulated by endothelial nitric oxide.

Recent clinical data suggest that subjects with sickle cell disease suffer from chronically impaired nitric oxide bioavailability. This has been attributed to increased consumption of nitric oxide by hemoglobin and reactive oxygen species, or decreased production of nitric oxide by endothelial cells; however the roles of nitric oxide bioavailability and endothelial dysfunction during acute pain crisis are controversial and incompletely understood. Although there have been several studies of endothelial function in steady state sickle cell disease, there has been no comprehensive study of endothelial function during pain crisis.

In this study, our primary objective is to measure the reactive hyperemia index (a measure of the endothelial response to shear stress) in twenty sickle cell subjects during acute pain crisis and to compare it with the reactive hyperemia index measured after recovery from pain crisis. This will identify whether there are acute changes in endothelial cell function during sickle cell pain crisis. Our secondary objective is to compare the reactive hyperemia index of thirty-five sickle cell subjects in steady state versus the reactive hyperemia index of thirty-five healthy control subjects. This will identify whether there are chronic differences in endothelial function between sickle cell subjects and healthy control subjects.

This study will determine if there are defects in endothelium-dependent vasodilation in response to shear stress during sickle cell pain crisis. Moreover, this study provides an opportunity to evaluate new physiologic biomarkers of sickle cell pain crisis based on measurements of blood flow, temperature, and oxygenation in the skin. These measurements may serve as clinical endpoints in future studies of disease pathogenesis or therapeutic interventions for sickle cell disease.

ELIGIBILITY:
* INCLUSION CRITERIA FOR SUBJECTS WITH SICKLE CELL DISEASE IN PAIN CRISIS:

  1. Age 18 years or older.
  2. Diagnosis of sickle cell anemia:

     1. Diagnosis of sickle cell disease (electrophoresis or HPLC documentation of hemoglobin SS, SC, S-beta-thalassemia or other hemoglobinopathies causing sickle cell disease is required).
     2. Acute onset pain crisis in a distribution typical for that subject, onset within the last 7 days and for which hospitalization and parenteral narcotic pain treatment are required.
  3. Ability to provide informed written consent.

EXCLUSION CRITERIA FOR SUBJECTS WITH SICKLE CELL DISEASE IN PAIN CRISIS:

1. Pregnancy.
2. History of non-trivial injury, burns, surgery or skin ulcers on the arms.
3. Carrier of drug resistant bacteria that normally requires isolation while visiting a hospital.
4. Administration of any of the following drugs within the last 14 days:

   * Phosphodiesterase-5 inhibitors (sildenafil, vardenafil, tadalafil)
   * Endothelin-1 receptor blockers (bosentan, sitaxentan, ambrisentan, tezosentan)
   * Nitric oxide donors (nitroglycerin, nitroprusside, nitrates)
5. Ingestion of caffeine within the 12 hours before the start of the study appointment, or tobacco use within the 30 days before the study appointment.
6. Diagnosis with any of the following chronic diseases or conditions:

   * Uncontrolled high blood pressure (systolic blood pressure must not be greater than 160 mmHg or diastolic blood pressure greater than 90 mmHg)
   * Uncontrolled high cholesterol (total cholesterol must not be greater than 240 mg/dL)
   * Uncontrolled diabetes (must not have both a documented history of diabetes and random blood glucose of greater than 200 mg/dL)
   * Chronic kidney disease (serum creatinine must not be greater than 2 mg/dL)
   * Coronary artery disease
   * Peripheral vascular disease
7. Received a blood transfusion within 7 days of the study procedure.

SICKLE CELL DISEASE SUBJECTS IN STEADY STATE

INCLUSION CRITERIA FOR SUBJECTS WITH SICKLE CELL DISEASE IN STEADY STATE:

1. Age 18 years or older.
2. Diagnosis of sickle cell anemia:

   a.Diagnosis of sickle cell disease (electrophoresis or HPLC documentation of hemoglobin SS, SC, S-beta-thalassemia or other hemoglobinopathies causing sickle cell disease is required).
3. Ability to provide informed written consent.

EXCLUSION CRITERIA FOR SUBJECTS WITH SICKLE CELL DISEASE IN STEADY STATE:

1. Pregnancy.
2. History of non-trivial trauma, burns, surgery or skin ulcers on the arms.
3. Carrier of drug resistant bacteria that normally requires isolation while visiting a hospital.
4. Experience of an acute pain crisis requiring intravenous (IV) narcotics and hospital admission within the last 14 days.
5. Ingestion of caffeine within the 12 hours before the start of the study appointment, or tobacco use within the 30 days before the study appointment.
6. Administration of any of the following drugs within the last 14 days:

   * Phosphodiesterase-5 inhibitors (sildenafil, vardenafil, tadalafil)
   * Endothelin-1 receptor blockers (bosentan, sitaxentan, ambrisentan, tezosentan)
   * Nitric oxide donors (nitroglycerin, nitroprusside, nitrates)
7. Diagnosis of any of the following chronic diseases or conditions: <TAB>

   * Uncontrolled high blood pressure (systolic blood pressure must not be greater than 160 mmHg or diastolic blood pressure greater than 90 mmHg)
   * Uncontrolled high cholesterol (total cholesterol must not be greater than 240 mg/dL)
   * Uncontrolled diabetes (must not have both a documented history of diabetes and random blood glucose of greater than 200 mg/dL)
   * Chronic kidney disease (serum creatinine must not be greater than 2 mg/dL)
   * Coronary artery disease
   * Peripheral vascular disease
8. Received a blood transfusion within 7 days of the study procedure.

HEALTHY CONTROL SUBJECTS

INCLUSION CRITERIA FOR HEALTHY CONTROL SUBJECTS

1. Age 18 years or older.
2. African, of African descent or Hispanic
3. Ability to provide informed written consent.

EXCLUSION CRITERIA FOR HEALTHY CONTROL SUBJECTS

1. Pregnancy.
2. History of non-trivial injury, burns, surgery or skin ulcers on the arms.
3. Carrier of drug resistant bacteria that normally requires isolation while visiting a hospital.
4. Administration of any of the following drugs within the last 14 days:

   * Phosphodiesterase-5 inhibitors (sildenafil, vardenafil, tadalafil)
   * Endothelin-1 receptor blockers (bosentan, sitaxentan, ambrisentan, tezosentan)
   * Nitric oxide donors (nitroglycerin, nitroprusside, nitrates)
5. Ingestion of caffeine in the 12 hours before the start of the study appointment, or used tobacco in the 30 days before the study appointment.
6. Diagnosis with any of the following chronic diseases or conditions:

   * Sickle cell disease <TAB>
   * Uncontrolled high blood pressure (systolic blood pressure must not be greater than 160 mmHg or diastolic blood pressure greater than 90 mmHg)
   * Uncontrolled high cholesterol (total cholesterol must not be greater than 240 mg/dL)
   * Uncontrolled diabetes (must not have both a documented history of diabetes and random blood glucose of greater than 200 mg/dL)
   * Chronic kidney disease (serum creatinine must not be greater than 2 mg/dL)
   * Coronary artery disease
   * Peripheral vascular disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2012-03-21; Study Completion 2018-10-05

SECONDARY OUTCOMES:
Skin Blood Flood | 1 month
Skin Temperature | 1 month
Tissue oxygenation | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Hans C Ackerman, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Platt OS, Thorington BD, Brambilla DJ, Milner PF, Rosse WF, Vichinsky E, Kinney TR. Pain in sickle cell disease. Rates and risk factors. N Engl J Med. 1991 Jul 4;325(1):11-6. doi: 10.1056/NEJM199107043250103. PMID 1710777
- [Background] Nagel RL. Sickle cell anemia is a multigene disease: sickle painful crises, a case in point. Am J Hematol. 1993 Jan;42(1):96-101. doi: 10.1002/ajh.2830420119. No abstract available. PMID 8416304
- [Background] Hebbel RP, Vercellotti GM. The endothelial biology of sickle cell disease. J Lab Clin Med. 1997 Mar;129(3):288-93. doi: 10.1016/s0022-2143(97)90176-1. No abstract available. PMID 9042813
- [Derived] Rowley CA, Ikeda AK, Seidel M, Anaebere TC, Antalek MD, Seamon C, Conrey AK, Mendelsohn L, Nichols J, Gorbach AM, Kato GJ, Ackerman H. Microvascular oxygen consumption during sickle cell pain crisis. Blood. 2014 May 15;123(20):3101-4. doi: 10.1182/blood-2013-11-533406. Epub 2014 Mar 24. PMID 24665133